CLINICAL TRIAL: NCT05836649
Title: Impact of Passive VR Versus Active VR on Heat Pain Thresholds and Pressure Pain Thresholds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Clinical Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 69330
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pain; Anxiety
Keywords: Thermal Sensory Analyzer (TSA-II); Peltier-Based Contact Thermode; Virtual Reality; Digital Algometer
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active VR then Passive VR (Experimental): Participant will conduct the Heat Pain Threshold experiment or Pressure Pain Threshold experiment using active VR first and then passive VR
  Interventions: Behavioral: Oculus Go headset without active intervention; Behavioral: Oculus Go headset with active intervention
- Passive VR then Active VR (Experimental): Participant will conduct the Heat Pain Threshold experiment or Pressure Pain Threshold experiment using passive VR first and then active VR
  Interventions: Behavioral: Oculus Go headset without active intervention; Behavioral: Oculus Go headset with active intervention
- No immersive virtual reality followed by immersive virtual reality (Experimental): Participant will conduct the Heat Pain Threshold experiment or Pressure Pain Threshold experiment using no immersive virtual reality first and then with immersive virtual reality.
  Interventions: Behavioral: Oculus Go headset without immersive virtual reality experience; Behavioral: Oculus Go headset with immersive virtual reality experience
- Immersive virtual reality followed by No immersive virtual reality (Experimental): Participant will conduct the Heat Pain Threshold experiment or Pressure Pain Threshold experiment using immersive virtual reality first and then with no immersive virtual reality.
  Interventions: Behavioral: Oculus Go headset without immersive virtual reality experience; Behavioral: Oculus Go headset with immersive virtual reality experience

INTERVENTIONS:
Behavioral: Oculus Go headset without active intervention — VR software with non-interactive content. Heat pain threshold (HPT) and pressure pain threshold (PPT) depends on the HPT limits test or PPT limits test.
  Arms: Active VR then Passive VR; Passive VR then Active VR
Behavioral: Oculus Go headset with active intervention — Participant will engage with the game display on the VR headset. Heat pain threshold (HPT) and pressure pain threshold (PPT) depends on the HPT limits test or PPT limits test.
  Arms: Active VR then Passive VR; Passive VR then Active VR
Behavioral: Oculus Go headset without immersive virtual reality experience — VR headset does not display any immersive virtual reality content. Heat pain threshold (HPT) and pressure pain threshold (PPT) depends on the HPT limits test or PPT limits test.
  Arms: Immersive virtual reality followed by No immersive virtual reality; No immersive virtual reality followed by immersive virtual reality
Behavioral: Oculus Go headset with immersive virtual reality experience — VR headset displays immersive virtual reality content. Heat pain threshold (HPT) and pressure pain threshold (PPT) depends on the HPT limits test or PPT limits test.
  Arms: Immersive virtual reality followed by No immersive virtual reality; No immersive virtual reality followed by immersive virtual reality

SUMMARY:
This is a prospective, crossover study of healthy participants evaluating the impact of passive vs. active virtual reality (VR) games on heat pain threshold (HPT) and pressure pain threshold (PPT).

DETAILED DESCRIPTION:
Virtual reality (VR) is an emerging, non-pharmaceutical intervention used to reduce perceived pain and anxiety in patients. VR's effect on pain and anxiety on patients is well-studied as is how VR games improve recalled pain and anxiety in pediatric burn and bone-fracture patients undergoing painful medical procedures. However, how differences in VR application construction (such as passive play vs. active play) impact patient perception of pain and anxiety is not well understood. In this study, we will measure the impact of passive vs. active VR applications on heat pain threshold (HPT) and pressure pain threshold (PPT), and immediate vs. recalled pain and anxiety levels.

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years of age
* English speaking
* hearing intact

Exclusion Criteria:

* a history of severe motion sickness
* currently have nausea
* history of seizures
* have hearing loss; are pregnant
* are currently taking beta blockers, chronotropic heart medications, or opioids or other prescription pain medications
* history of chronic pain or acute pain syndromes.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Change in heat pain threshold | Duration of intervention, approximately 15 minutes
  Heat pain threshold measured by the TSA Air II device. Temperature ranges from 32 degrees C to 50 degrees C, with higher temperatures indicating a higher heat pain threshold.

SECONDARY OUTCOMES:
Change in pressure pain threshold | Duration of intervention, approximately 15 minutes
  Pressure pain threshold measured by a computerized pressure pain algometer. Pressure ranges from 0 kPa to 1000 kPa, with higher pressures indicating a higher pressure pain threshold.
Change in recalled pain level | immediately after intervention, 24 hours after the intervention
  Recalled pain level measured by a numerical rating scale (NRS) from 0-10. Scale ranges from 0-10, with higher scores indicating higher pain levels.
Change in lower recalled fear/anxiety level | immediately after intervention, 24 hours after the intervention
  Fear/anxiety level measure by the anxiety scale. This scale ranges from 0-10, 0 meaning no anxiety and 10 indicating extreme or worst-possible anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Lucile Parkard Children's Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le May S, Hupin M, Khadra C, Ballard A, Paquin D, Beaudin M, Bouchard S, Cotes-Turpin C, Noel M, Guingo E, Hoffman HG, Dery J, Hung N, Perreault I. Decreasing Pain and Fear in Medical Procedures with a Pediatric Population (DREAM): A Pilot Randomized Within-Subject Trial. Pain Manag Nurs. 2021 Apr;22(2):191-197. doi: 10.1016/j.pmn.2020.10.002. Epub 2021 Jan 22. PMID 33495093
- [Background] Rolke R, Baron R, Maier C, Tolle TR, Treede -DR, Beyer A, Binder A, Birbaumer N, Birklein F, Botefur IC, Braune S, Flor H, Huge V, Klug R, Landwehrmeyer GB, Magerl W, Maihofner C, Rolko C, Schaub C, Scherens A, Sprenger T, Valet M, Wasserka B. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): standardized protocol and reference values. Pain. 2006 Aug;123(3):231-243. doi: 10.1016/j.pain.2006.01.041. Epub 2006 May 11. PMID 16697110
- [Background] Price J, Sloman L, Gardner R Jr, Gilbert P, Rohde P. The social competition hypothesis of depression. Br J Psychiatry. 1994 Mar;164(3):309-15. doi: 10.1192/bjp.164.3.309. PMID 8199784
- [Derived] Rodriguez ST, Jimenez RT, Wang EY, Zuniga-Hernandez M, Titzler J, Jackson C, Suen MY, Yamaguchi C, Ko B, Kong JT, Caruso TJ. Virtual reality improves pain threshold and recall in healthy adults: A randomized, crossover study. J Clin Anesth. 2025 Apr;103:111816. doi: 10.1016/j.jclinane.2025.111816. Epub 2025 Mar 21. PMID 40117909